CLINICAL TRIAL: NCT05615831
Title: The Impact of Exercise With Blood Flow Restriction: Sex and Age Differences on Physical Performance, Muscle Hypertrophy, and Blood Biomarkers
Brief Title: The Impact of Exercise With Blood Flow Restriction: Sex and Age Differences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Brunswick (Other)
Collaborators: Public Health Agency of Canada (PHAC) (Other Government)
Responsible Party: Principal Investigator, Martin Senechal, Associate Professor, Martin Senechal, Ph.D., University of New Brunswick
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021-124
Record Dates: First submitted 2022-09-20; First posted 2022-11-14 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Physical Activity
Keywords: Blood flow restriction; Sex comparisons; Resistance training; Sex Differences; Aging; Young healthy; Strength Training
MeSH Terms: conditions — Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Young adult (19-30 years) (Experimental): Individuals aged 19-30 who are not physically active will participate in resistance training combined with blood flow restriction.
  Interventions: Behavioral: Resistance Training with Blood flow restriction
- Older adults adult (aged 65 years and older) (Experimental): Individuals aged 65 years and older who are not physically active will participate in resistance training combined with blood flow restriction.
  Interventions: Behavioral: Resistance Training with Blood flow restriction

INTERVENTIONS:
Behavioral: Resistance Training with Blood flow restriction — Participants will perform six weeks of blood flow restriction (60% occlusion) combined with resistance training at 30% of 1RM. The intervention comprises five exercises: incline chest press, seated row, leg press, knee extension, and knee flexion. The protocol is as follows: 30 repetitions followed by three sets of 15 repetitions for a total of four sets and 75 repetitions per exercise. There will be a one-minute recovery between sets where the cuffs remain inflated and a four-minute recovery between exercises where the cuffs will be deflated.

SUMMARY:
The primary objective is to investigate whether six weeks of resistance training, in combination with blood flow restriction, produces a different adaptation in fat-free mass between males and females that are not physically active. The secondary objective is to compare changes in physical function, physical performance, and blood biomarkers between males and females following resistance training and blood flow restriction.

DETAILED DESCRIPTION:
Previous studies indicated a reduced workload (i.e., lifting lighter weight) combined with blood flow restriction leads to increased fat-free mass and muscle strength. However, females have been underrepresented in the blood flow restriction literature. Therefore, no study has investigated whether males and females of different age groups have different adaptations in fat-free mass, muscle strength, and performance outcomes following resistance training using blood flow restriction.

The primary objective will be to investigate sex differences in fat-free mass following six weeks of resistance training combined with blood flow restriction in young and older adults.

The secondary objective is to investigate sex differences in muscle strength, physical performance, and blood biomarkers between males and females following resistance training and blood flow restriction.

Briefly, participants between 19-30 years and 65 years and older will be recruited to participate in this study. Participants will present to the laboratory for two baseline testing visits interspersed with a minimum of four days. The first testing visit will include a variety of questionnaires, a blood draw, lipid and glucose, a dual-energy x-ray absorptiometry scan, anthropometrics, and a submaximal VO2. The second visit will include several physical function tests, such as the short physical performance battery and the Y-balance test, as well as a high-intensity isokinetic fatigue test using isokinetic dynamometry and 1-repetition maximum testing.

Upon completion of baseline testing, participants are enrolled in the exercise program. The first exercise session includes a blood draw before and immediately after the training session. This procedure will be duplicated at the final exercise session at the end of the six weeks.

Participants' full occlusion will be estimated using the formula developed by Loenneke et al. (2015). Then each participant's occlusion will be set at 60% of each individual's total limb occlusion. This will be used in combination with the following exercises incline chest press, seated row, leg press, knee extension, and knee flexion performed at 30% of 1RM. The protocol is as follows: 30 repetitions followed by three sets of 15 repetitions for a total of four sets and 75 repetitions per exercise. There will be a one-minute recovery between sets where the cuffs remain inflated and a four-minute recovery between exercises where the cuffs will be deflated.

Following the completion of the six weeks of exercise, participants will again present to the laboratory for two follow-up visits similar to the first two baseline visits.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 19 and 100 years
* Sedentary (not meeting physical activity guidelines), but otherwise healthy

Exclusion Criteria:

* Aged outside the threshold
* Uncontrolled hypertension
* Presence of cardiovascular disease
* Either surgery, bone fracture, or skin graft within the previous three months
* Uncontrolled diabetes mellitus
* Pregnancy
* Individuals taking medications known to increase risk of blood clotting

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
Muscle hypertrophy | Baseline and 6 weeks
  Change in fat-free mass

SECONDARY OUTCOMES:
Strength | Baseline and 6 weeks
  Change in 1-repetition maximum
Muscle Power | Baseline and 6 weeks
  Change in vertical jump score
Muscle Endurance | Baseline and 6 weeks
  Change in knee extension and flexion
Changes in physical function | Baseline and 6 weeks
  Changes in short physical performance battery, senior fitness test, and Y-balance test
Changes in blood biomarkers | Baseline and 6 weeks post-intervention and pre and post an acute bout of resistance training at baseline and and after 6 weeks
  Changes in circulating blood biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Martin Senechal, PhD, Principal Investigator — University of New Brunswick
Locations (1):
- University of New Brunswick - Kinesiology, Fredericton, New Brunswick, Canada

REFERENCES:
- [Derived] Arnason JK, Thomson AM, Peskett LE, Nancekievill DA, Bouchard DR, Senechal M. Age-Related Differences in Adaptation of Lean Body Mass, Muscle Strength, and Performance Following 6 Weeks of Blood Flow Restriction Training in Young and Older Adults. J Frailty Sarcopenia Falls. 2025 Mar 1;10(1):37-47. doi: 10.22540/JFSF-10-037. eCollection 2025 Mar. PMID 40035085